CLINICAL TRIAL: NCT06934083
Title: A Novel Family E-Health Intervention Process To Reduce Childhood Obesity
Brief Title: Lifestyle Medicine Health Education and Intervention Program "Family Central E-Health"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Texas Health Science Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RF00187; 2U54MD006882-06 (NIH)
Record Dates: First submitted 2021-09-28; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Life Style, Healthy; Behavioral Changes
Keywords: obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: This randomized control study will examine knowledge, attitudes, and healthy lifestyle practices regarding six "Lifestyle Medicine Health Education" topics among caregivers of Pediatric patients. In addition, clinical outcomes such as blood pressure, blood glucose, total cholesterol, waist circumference, and Body Mass Index (BMI) will be assessed; and the study will assess the change in outcomes from baseline to completion of this program. After enrollment, the study team will deliver a scale and a tape measure to the caregiver at the address of their choice. The participants' biometric measurements will be submitted via our text-messaging platform. Participants will be assigned into one of two research arms a) the e-health intervention group or b) a control group of usual care. All participants will engage in the study with non-web- based, two-way text messaging via their personal cell phone.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-health education briefs (Experimental): The e-health intervention group will receive health education briefs that will cover all six lifestyle modifications every 6 weeks. Over the 6-month study period, each lifestyle modification topic will be covered 4 times.
  Interventions: Behavioral: E-health education briefs
- Usual care (No Intervention): The usual care group will receive text messages directing caregivers to consult the electronic medical record patient portal of their child, which has a library of health literature, related to lifestyle behaviors, their child's lab results, and appointment reminders.

INTERVENTIONS:
Behavioral: E-health education briefs — Participants will be asked to complete self-administered questionnaire regarding the six healthy lifestyles delivered via text message to their cell phone. Then, during the six-month intervention, participants will receive text messages at intervals set by their preference but at least 2 times per week to ensure adequate space for education delivery and assessment through Likert scale text message surveys relating to Lifestyle Health Education topics including Nutrition, Physical Activity, Tobacco Avoidance, Sleep, Stress Management, and Social Connection. As to the clinical outcomes, self-reported blood pressure, blood glucose, total cholesterol, waist circumference, and body mass index (BMI) will be collected from the participants at enrollment and at the live or virtual community celebration at the close of the study.
  Arms: E-health education briefs

SUMMARY:
Participants will receive text messages at intervals set by preference but at least 2 times per week relating to Lifestyle Health Education for 6 months. The topics to be reviewed include: Nutrition, Physical Activity, Tobacco Avoidance, Sleep, Stress Management, and Social Connection. Participants will be asked to complete surveys regarding these topics at the beginning and end of the week; in addition, participants will self report to the study team vital signs (including blood pressure, blood glucose, total cholesterol, waist circumference, and body mass index (BMI)) at the beginning and end of the study. Although there is a chance participants may encounter some issues with the study procedures (possible breach of confidentiality, or issues with the study procedures), these risks are minimal. The study team will always keep information secure, and participants may decline to participate in any study procedures, or withdraw from the study, at any time.

One benefit from this study may be that participants may improve their overall health by learning more about healthy eating, improved physical activity, limiting/avoiding tobacco intake, improved sleep patterns, adequate stress management, and better social connection. Participation in this study is not required.

DETAILED DESCRIPTION:
Participants will be randomized (like the flip of coin) to one of two study groups. Based on the group assigned, participants will receive text messages which include either: 1) reminders of health education available through the patient portal of the electronic medical record for participant's child, or 2) briefs on six health education topics: nutrition, physical activity, sleep, tobacco avoidance, stress management, and social connection. No matter which group assigned, participants will attend one live or virtual group meeting to close the study.

For both groups, researchers will measure knowledge, attitudes and health habits before and after the program. Researchers will also request self-reports of health status (height, weight, waist size, Body Mass Index (BMI), blood pressure, blood sugar, and total cholesterol). Participants will provide the researchers with estimates of most recent blood pressure, total cholesterol, and blood glucose test if known. The study will include text message briefs received at least twice weekly for six months, and will include the following measures:

* General information (e.g., age, gender, education)
* Health knowledge & attitudes (e.g., heart disease, diabetes) & healthy lifestyle practices (e.g., diet, exercise)
* Health status (e.g., Blood pressure, BMI, etc.) The study team estimate that 142 people will enroll in the study.

For both groups, the following will be measured at the first visit (also called the "baseline visit" completed at the time of enrollment) and also at the last visit (during the live or virtual community celebration):

* Participant's health status (height, weight, waist size, Body Mass Index (BMI), blood pressure, blood sugar, and total cholesterol).
* Survey of knowledge, attitudes and health habits.

As described above, participants will be randomized to one of two groups:

1. If selected to be in the first group, participants will first receive a welcome text with a link to the patient portal for the electronic health record (of participant's child). Participants will then receive weekly reminders of health education (one reminder each week for 6 months), available through the patient portal of the electronic medical record (of participant's child). At least twice a week, participants will also complete surveys regarding participant's knowledge, attitudes and behaviors of the health education topics (these surveys will be delivered to their phone via text messages).
2. If selected to be in the second group, participants will begin receiving weekly text messages which include health education briefs on 6 different topics (one text message a week for 6 months). At least twice a week, participants will also complete surveys regarding participants' knowledge, attitudes and behaviors of the health education topics (these surveys will be delivered to participant's phone via text messages).

ELIGIBILITY:
Inclusion Criteria:

* family member has a child who is a current or former patient of Pediatric Mobile Clinic with a medical diagnosis of overweight/obese,
* defined as BMI percentile of 85% or above,
* age of the child is 6 months to 11 years old,
* family member is a primary caregiver to the child,
* family member over the age of 18 years,
* family member is not currently pregnant, and
* family member has a cell phone with Short Message Service (SMS) text message capability.

Exclusion Criteria:

* family member has a terminal illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Motivation in units of scale measure | 12 months
  10-point Likert scale (minimum of 1, maximum of 10, 10 representing highest level of motivation) of transtheoretical stage of change used to assess motivation to achieve participant derived SMART goal each week for 6 months then at 3-month intervals for 2 follow-up check-ins.

SECONDARY OUTCOMES:
Confidence in units of scale measure | 12 months
  10-point Likert scale (minimum of 1, maximum of 10, 10 representing highest level of confidence) of transtheoretical stage of change used to assess confidence to achieve participant derived SMART goal each week for 6 months then at 3-month intervals for 2 follow-up check-ins.

OTHER OUTCOMES:
SMART goal | 12 months
  Participant created goal that is specific, measurable, achievable, and time bound. Goal is related to lifestyle behavior modifications with assessment of achievement each week for 6 months then assessed at 3-month intervals for 6 following months. This is qualitative data that has no minimum, maximum, or standardization of better vs. worse.
BMI in kg/m^2 | 6 months
  self-reported body weight using provided weight scale and self-reported recall height
Total Cholesterol in milligrams (mg) of cholesterol per deciliter (dL) of blood | 6 months
  self reported recall of cholesterol level
Blood glucose in mg/dl (milligrams per deciliter) | 6 months
  self reported recall of blood sugar either from venipuncture or capillary stick
Blood pressure in millimeters of mercury (mmHg) | 6 months
  self-reported recall of automated or manual systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Christina Robinson, MD, Principal Investigator — UNTHSC
Locations (1):
- UNT Health Science Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No
All study-related materials and documentation will only be accessible to the study personnel. Completed questionnaires will be placed into locked file cabinets in the office of the PI. Clinical outcomes recorded through a shared Microsoft excel drive will only be accessible to key study personnel.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study protocol documents (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT06934083/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Cover page (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/83/NCT06934083/Prot_SAP_001.pdf